CLINICAL TRIAL: NCT03448692
Title: A PHASE 2, 24-WEEK, ADAPTIVE, OPEN LABEL, SEQUENTIAL COHORT TRIAL TO EVALUATE THE EFFICACY, SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF-06730512 FOLLOWING MULTIPLE DOSES IN ADULT SUBJECTS WITH FOCAL SEGMENTAL GLOMERULOSCLEROSIS (FSGS)
Brief Title: A Study to Evaluate PF-06730512 in Adults With Focal Segmental Glomerulosclerosis (FSGS)
Acronym: PODO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of efficacy at both tested doses on 5th December 2022. The decision to terminate the study is not related to a safety concern.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: C0221002; 2019-003607-35 (EudraCT Number); ROBO2 (Other: Alias Study Number); PODO (Other: Alias Study Number)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Focal Segmental Glomerulosclerosis (FSGS)
Keywords: Proteinuria
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Proteinuria | interventions — PF-06730512

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-06730512 Cohort 1 (Experimental): Subjects in cohort 1 will receive dose 1 Intravenous (IV) infusion.
  Interventions: Drug: PF-06730512
- PF-06730512 Cohort 2 (Experimental): Subjects in cohort 2 will receive dose 2 IV infusion.
  Interventions: Drug: PF-06730512
- PF-06730512 Cohort 3 (optional) (Experimental): Subjects in cohort 3 will receive dose 3 IV infusion.
  Interventions: Drug: PF-06730512

INTERVENTIONS:
Drug: PF-06730512 — Subjects in cohort 1 will receive Dose 1 Intravenous infusion (IV). Subjects in cohort 2 will receive Dose 2 IV. Subjects in cohort 3 will receive Dose 3 IV infusion.

SUMMARY:
The purpose of this Phase 2 adaptive study is to evaluate the efficacy, safety, tolerability and pharmacokinetics of PF-06730512 following multiple intravenous infusions in adult subjects with FSGS.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 years and older who have a confirmed biopsy diagnosis of FSGS.
2. Estimated glomerular filtration rate (eGFR) greater than or equal to 45 ml/min/1.73 m2. If eGFR is 30 - 45 ml/min/1.73 m2, a recent biopsy (within 12 months prior to Screening) must demonstrate < 50% tubulointerstitial fibrosis.
3. Urine protein:creatinine ratio (UPCR) greater than 1.5 g/g at screening.
4. Treated with at least one but not more than 3 classes of immunosuppressants either alone or in combination, or has a contraindication to use of an immunosuppressant or is intolerant to an immunosuppressant per investigator judgment.

Exclusion Criteria:

1. Diagnosis of collapsing FSGS.
2. Advanced chronic changes on renal biopsy as evidenced by greater than 50% tubulointerstitial fibrosis.
3. Organ transplant.
4. History of malignancy, with the exception of basal or squamous cell carcinoma that has been treated and fully resolved for a minimum of 5 years.
5. Body mass index (BMI) greater than 45 kg/m2.
6. Subjects with a history of prior treatment with or use of interferon, lithium, pamidronate, mTOR inhibitors (eg, sirolimus), testosterone/anabolic steroids, anthracycline (eg, doxorubicin), heroin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (108):
- United States (56):
  - The Kirklin Clinic of University Alabama Birmingham Hospital, Birmingham, Alabama
  - Investigational Drug Service Pharmacy UAB Hosptial, Birmingham, Alabama
  - Clinical Research Unit at UAB Hospital, Birmingham, Alabama
  - UAB Nephrology Research Clinic at Paula Building, Birmingham, Alabama
  - Academic Medical Research Institute, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Cedars-Sinai Ambulatory Infusion Center, Los Angeles, California
  - Cedars-Sinai Comprehensive Transplant Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Clinical and Translational Research Center, Los Angeles, California
  - UCLA Department of Medicine, Los Angeles, California
  - Clinical and Translation Research Unit, Palo Alto, California
  - Stanford University-Nephrology Division, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Stanford Health Care Investigational Pharmacy, Stanford, California
  - Stanford University-Nephrology Division, Stanford, California
  - Stanford University, Stanford, California
  - Yale Center for Clinical Investigation Hospital Research Unit, New Haven, Connecticut
  - Yale Nephrology Clinical Research Clinic, New Haven, Connecticut
  - Yale University School of Medicine - Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale Center for Clinical Investigation - Church Street Research Unit, New Haven, Connecticut
  - University of Miami Hospital and Clinics, Miami, Florida
  - University of Miami Katz Family Division of Nephrology, Miami, Florida
  - University of Miami, Miami, Florida
  - Georgia Nephrology Research Institute, Lawrenceville, Georgia
  - Georgia Nephrology, Lawrenceville, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johnson County Clin Trials, Lenexa, Kansas
  - Boston Medical Center - Interventional Radiology, Boston, Massachusetts
  - Boston Medical Center - Nephrology, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Boston University - GCRU, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - St. Luke's Hospital, Kansas City, Missouri
  - New York University Grossman School of Medicine - CTSI, New York, New York
  - UNC Eastowne, Chapel Hill, North Carolina
  - UNC Clinical and Translational Research Center, Chapel Hill, North Carolina
  - University of Cincinnati at DCI McMillan Research Unit, Cincinnati, Ohio
  - Hoxworth Center Subspecialties Clinic, Cincinnati, Ohio
  - UC Health Barrett Center, Cincinnati, Ohio
  - UC Health Medical Arts Building, Cincinnati, Ohio
  - University of Cincinnati Gardner Neuroscience Institute, Cincinnati, Ohio
  - The Cleveland Clinic - Investigational Drug Pharmacy, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - CarePoint East at The Ohio State University, Columbus, Ohio
  - The Ohio State University Clinical Research Center, Columbus, Ohio
  - The Ohio State University Investigational Drug Services, Columbus, Ohio
  - The Ohio State University Wexner Medical Center- Nephrology Clinical Trials Unit, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Kidney and Hypertension Care Center, PA, Houston, Texas
  - Southside Pharmacy, Houston, Texas
  - Prolato Clinical Research Center (PCRC), Houston, Texas
  - Baylor Scott & White Clinic - Temple South Loop, Temple, Texas
- Canada (11):
  - University of Alberta - Pharmacy Research Office, Edmonton, Alberta
  - University of Alberta - Clinical Investigation Unit, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Pacific Nephrology Group, Vancouver, British Columbia
  - Vancouver General Hospital/Vancouver Coastal Health, Vancouver, British Columbia
  - St. Paul's Hospital/Providence Health Care, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre - Kidney Care Centre at the CNIB, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CIUSSS de l'Est-de-l'Ile-de-Montreal - installation Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre for Innovative Medicine, Research Institute of the McGill University Health Centre, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (3):
  - Hopital Henri Mondor, Créteil
  - CHU de Nice - Hopital Pasteur, Nice
  - Hopital Necker - Enfants Malades, Paris
- Germany (9):
  - Universitätsklinikum Dresden, Medizinische Klinik III, Nephrologie, Dresden, Saxony
  - Universitaetsklinikum Aachen, Aachen
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Uniklinik Koeln, Cologne
  - Universitaetsklinikum Erlangen, Erlangen
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Mannheim, Mannheim
  - Nephrologisches Zentrum Villingen-Schwenningen, Villingen-Schwenningen
  - Sidonia Apotheke, Villingen-Schwenningen
- Italy (2):
  - Ics Maugeri Spa-Sb Irccs, Pavia PV, Pavia
  - Asst Papa Giovanni Xxiii, Bergamo
- Japan (5):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka University Hospital, Suita, Osaka
  - National Hospital Organization Chiba-East Hospital, Chiba
  - Niigata University Medical & Dental Hospital, Niigata
- Mexico (3):
  - Hospital Universitario "Dr Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - SMIQ S de RL de CV, Querétaro
- Poland (4):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Lodz
  - Apteka Szpitalna SPZOZ, Lodz
  - Centrum Zdrowia MDM, Warsaw
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw
- Slovakia (3):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Bratislava
  - Narodny ustav detskych chorob, Bratislava
- Spain (4):
  - Hospital Público Da Mariña, Burela de Cabo, LUGO
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (6):
  - Oxford University Hospitals NHS Foundation Trust, Headington, Oxford
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry
  - St. George's University Hospitals NHS Foundation Trust, London
  - Hammersmith Hospital, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Beck LH Jr, Berasi SP, Copley JB, Gorman D, Levy DI, Lim CN, Henderson JM, Salant DJ, Lu W. PODO: Trial Design: Phase 2 Study of PF-06730512 in Focal Segmental Glomerulosclerosis. Kidney Int Rep. 2021 Apr 3;6(6):1629-1633. doi: 10.1016/j.ekir.2021.03.892. eCollection 2021 Jun. PMID 34169203
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0221002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 47 participants were enrolled into the study. All participants received treatment.
Groups:
- PF-06730512 1000 mg IV: Participants received PF-06730512 1000 milligram (mg) intravenously (IV) every 2 weeks (Q2W).
- PF-06730512 300 mg IV: Participants received PF-06730512 300 mg IV Q2W.
Period: Disposition Phase:Screening:up to 43Days
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0
Period: Lead in Period:8 Weeks (W)
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Started | 23 | 24
Completed | 23 | 24
Not Completed | 0 | 0
Period: Investigational Treatment Period:Upto24W
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Started | 23 | 24
Completed | 22 | 15
Not Completed | 1 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician's decision | 0 | 1
Not completed — Study terminated by sponsor | 0 | 5
Not completed — Withdrawal by Subject | 0 | 2
Period: Follow up Period:9 Weeks
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Started | 23 (Participants who discontinued treatment period also entered follow up period.) | 23 (Participants who discontinued treatment period also entered follow up period.)
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) was defined as all enrolled participants who had received at least one dose of study treatment.
Groups:
- PF-06730512 1000 mg IV: Participants received PF-06730512 1000 mg IV Q2W.
- Total: Total of all reporting groups
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (13.64) | 41.0 (14.60) | 41.8 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 11 | 14 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 18 | 21 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 20 | 16 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Urinary Protein to Creatinine Ratio (UPCR) Based on 24-hour Urine Collection at Week 13
Description: UPCR is a ratio between two measured substances in urine: milligram of protein per millimole (mmol) of creatinine, reported in units mg/mmol. A decrease in UPCR may be associated with improved renal and cardiovascular function.
Time Frame: Baseline, Week 13
Population: The Full Analysis Set (FAS) was defined as all enrolled participants who had received at least one dose of study treatment and had at least one post-baseline measurement of UPCR based on 24-hour urine collection. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 21 | 19
Percentage change | -12.283 [-26.096 to 4.112] | -0.045 [-9.528 to 10.432]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event was considered treatment emergent relative to a given treatment if the event occurred for the first time during the investigational treatment period and was not seen prior to the start of treatment (during the lead-in period), or the event was seen prior to the start of treatment but increased in severity during treatment. Adverse events occurring during the lead-in period were considered non-treatment emergent. Events that occurred during the follow-Up period were counted as treatment emergent and attributed to the previous treatment taken.
Time Frame: From Day 1 of treatment up to 9 weeks after last dose of study treatment (up to Week 33)
Population: SAS was defined as all enrolled participants who had received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Participants | 20 | 17

3. Secondary Outcome: Number of Participants With Abnormalities in Laboratory Test Parameters
Description: Hemoglobin (Hg), hematocrit, erythrocytes: <0.8*lower limits of normal (LLN); platelets: <0.5*LLN>1.75*upper limits of normal(ULN); leukocytes (leu), glucose-fasting:<0.6*LLN>1.5*ULN; lymphocytes (lym), lym/leu, neutrophils(neu),neu/leu, protein, albumin, phosphate, free thyroxine, thyroid stimulating hormone: <0.8*LLN>1.2*ULN; basophils (bas), bas/leu, eosinophils (eos), eos/leu, monocytes(mon), mon/leu: >1.2*ULN; bilirubin (total, direct, indirect):>1.5*ULN; aspartate aminotransferase(AT), alanine AT, lactate dehydrogenase, alkaline phosphatase:>3.0*ULN; blood urea nitrogen, creatinine, cholesterol (total,LDL,HDL),triglycerides, Hg A1C: >1.3*ULN; sodium: <0.95*LLN>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate: <0.9*LLLN>1.1*ULN; prolactin: >1.1*ULN; creatine kinase: >2.0*ULN; urobilinogen: >=1; Urine-specific gravity: <1.003>1.030, pH: <4.5 >8, glucose,protein,bilirubin,nitrite,leukocyte esterase, ketones: >=1.Categories with at-least 1 non-zero values are reported.
Time Frame: From Day 1 of treatment up to Week 33
Population: SAS was defined as all enrolled participants who had received at least one dose of study treatment. Here, 'Number Analyzed' signifies number of participants evaluable for the specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Participants
  Hematology: Hemoglobin < 0.8 * Lower Limit Number (LLN) | 5 | 4
  Hematology: Hematocrit < 0.8 * LLN | 5 | 7
  Hematology: Erythrocytes < 0.8 * LLN | 3 | 4
  Hematology: Ery. Mean Corpuscular Volume < 0.9 * LLN | 1 | 0
  Hematology: Ery. Mean Corpuscular Hemoglobin < 0.9 * LLN | 1 | 0
  Hematology: Platelets> 1.75 * ULN | 1 | 0
  Hematology: Lymphocytes< 0.8 * LLN | 0 | 4
  Hematology: Lymphocytes/Leukocytes < 0.8 * LLN | 1 | 6
  Hematology: Lymphocytes/Leukocytes > 1.2 * ULN | 0 | 1
  Hematology: Neutrophils < 0.8 * LLN | 1 | 2
  Hematology: Neutrophils > 1.2 * ULN | 3 | 4
  Hematology: Neutrophils/Leukocytes < 0.8 * LLN | 1 | 1
  Hematology: Neutrophils/Leukocytes > 1.2 * ULN | 0 | 1
  Hematology: Eosinophils > 1.2 * ULN | 2 | 1
  Hematology: Eosinophils/Leukocytes> 1.2 * ULN | 3 | 3
  Hematology: Monocytes/Leukocytes> 1.2 * ULN | 0 | 1
  Clinical chemistry: Aspartate Aminotransferase > 3.0 * ULN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Aspartate Aminotransferase > 3.0 * ULN | 1 | 0
  Clinical chemistry: Alanine Aminotransferase > 3.0 * ULN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Alanine Aminotransferase > 3.0 * ULN | 1 | 0
  Clinical chemistry: Protein < 0.8 * LLN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Protein < 0.8 * LLN | 9 | 11
  Clinical chemistry: Albumin < 0.8 * LLN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Albumin < 0.8 * LLN | 8 | 11
  Clinical chemistry: Blood Urea Nitrogen > 1.3 * ULN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Blood Urea Nitrogen > 1.3 * ULN | 10 | 8
  Clinical chemistry: Creatinine > 1.3 * ULN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Creatinine > 1.3 * ULN | 8 | 12
  Clinical chemistry: Urate > 1.2 * ULN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Urate > 1.2 * ULN | 3 | 2
  Clinical chemistry: Cholesterol > 1.3 * ULN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Cholesterol > 1.3 * ULN | 6 | 7
  Clinical chemistry: HDL Cholesterol < 0.8 * LLN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: HDL Cholesterol < 0.8 * LLN | 1 | 0
  Clinical chemistry: LDL Cholesterol > 1.2 * ULN: number analyzed (Participants) | 23 | 22
  Clinical chemistry: LDL Cholesterol > 1.2 * ULN | 6 | 5
  Clinical chemistry: Triglycerides > 1.3 * ULN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Triglycerides > 1.3 * ULN | 6 | 8
  Clinical chemistry: Sodium < 0.95 * LLN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Sodium < 0.95 * LLN | 1 | 0
  Clinical chemistry: Potassium < 0.9 * LLN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Potassium < 0.9 * LLN | 1 | 0
  Clinical chemistry: Potassium > 1.1 * ULN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Potassium > 1.1 * ULN | 1 | 0
  Clinical chemistry: Calcium < 0.9 * LLN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Calcium < 0.9 * LLN | 1 | 3
  Clinical chemistry: Bicarbonate < 0.9 * LLN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Bicarbonate < 0.9 * LLN | 0 | 1
  Clinical chemistry: Glucose > 1.5 * ULN: number analyzed (Participants) | 23 | 23
  Clinical chemistry: Glucose > 1.5 * ULN | 2 | 2
  Urinalysis: Specific Gravity > 1.030: number analyzed (Participants) | 21 | 24
  Urinalysis: Specific Gravity > 1.030 | 5 | 6
  Urinalysis: pH > 8 | 1 | 0
  Urinalysis: Urine Glucose >= 1 | 5 | 10
  Urinalysis: Urine Protein >=1 | 22 | 24
  Urinalysis: Urine Hemoglobin >=1 | 15 | 17
  Urinalysis: Nitrite >= 1 | 1 | 3
  Urinalysis: Leukocyte Esterase >= 1 | 5 | 6
  Urinalysis: Urine Erythrocytes >= 20: number analyzed (Participants) | 22 | 24
  Urinalysis: Urine Erythrocytes >= 20 | 3 | 3
  Urinalysis: Urine Leukocytes >= 20: number analyzed (Participants) | 22 | 24
  Urinalysis: Urine Leukocytes >= 20 | 2 | 5
  Urinalysis: Granular Casts > 1: number analyzed (Participants) | 5 | 2
  Urinalysis: Granular Casts > 1 | 4 | 2
  Urinalysis: Hyaline Casts > 1: number analyzed (Participants) | 18 | 18
  Urinalysis: Hyaline Casts > 1 | 17 | 15
  Urinalysis: Urine Creatinine <40 | 9 | 8
  Urinalysis: Urine Creatinine >300 | 1 | 0
  Urinalysis: Urine (24HR) Creatinine > 1.1 * ULN | 2 | 6

4. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight and at baseline values were reported for this outcome measure.
Time Frame: Baseline, Change at Weeks 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 33
Population: SAS was defined as all enrolled participants who had received at least one dose of study treatment. Here, 'Number Analyzed' signifies number of participants evaluable for the specific timepoints.
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Kilogram
  Baseline | 78.3 (17.8) | 88.9 (23.5)
  Week 2 | 1.0 (2.2) | -0.3 (1.9)
  Week 3: number analyzed (Participants) | 23 | 23
  Week 3 | 0.4 (2.5) | -0.3 (2.2)
  Week 5: number analyzed (Participants) | 22 | 23
  Week 5 | 0.5 (3.0) | -0.5 (4.8)
  Week 7: number analyzed (Participants) | 23 | 22
  Week 7 | 0.6 (2.6) | -1.0 (5.3)
  Week 9: number analyzed (Participants) | 22 | 22
  Week 9 | 0.1 (3.1) | -0.4 (3.4)
  Week 11: number analyzed (Participants) | 22 | 20
  Week 11 | 0.7 (2.8) | -0.1 (4.2)
  Week 13: number analyzed (Participants) | 23 | 22
  Week 13 | -0.2 (1.9) | -1.0 (3.4)
  Week15: number analyzed (Participants) | 4 | 13
  Week15 | -0.3 (1.0) | -0.7 (4.0)
  Week 17: number analyzed (Participants) | 4 | 9
  Week 17 | -0.2 (1.2) | -1.2 (4.8)
  Week 19: number analyzed (Participants) | 4 | 9
  Week 19 | -0.4 (1.0) | -1.3 (4.8)
  Week 21: number analyzed (Participants) | 4 | 9
  Week 21 | 0.3 (1.7) | -1.3 (4.9)
  Week 23: number analyzed (Participants) | 4 | 9
  Week 23 | 0.3 (1.2) | -1.5 (5.3)
  Week 25: number analyzed (Participants) | 4 | 16
  Week 25 | -0.1 (1.6) | -1.1 (4.8)
  Week 27: number analyzed (Participants) | 4 | 16
  Week 27 | 0.7 (1.4) | -0.6 (5.2)
  Week 29: number analyzed (Participants) | 4 | 16
  Week 29 | 0.5 (1.5) | -1.0 (4.5)
  Week 33: number analyzed (Participants) | 4 | 16
  Week 33 | 0.5 (1.6) | -0.6 (5.4)

5. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Change from baseline in blood pressure and at baseline values were reported for this outcome measure.
Time Frame: Baseline, Change at Weeks 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 33
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Millimeter of mercury (mmHg)
  Baseline | 131.2 (12.8) | 125.3 (11.8)
  Week 2 | -1.8 (13.1) | -1.3 (7.8)
  Week 3: number analyzed (Participants) | 23 | 23
  Week 3 | -1.3 (10.2) | 1.7 (7.5)
  Week 5: number analyzed (Participants) | 22 | 23
  Week 5 | -3.0 (10.6) | -1.9 (9.0)
  Week 7: number analyzed (Participants) | 23 | 22
  Week 7 | -2.0 (11.3) | -1.2 (9.0)
  Week 9: number analyzed (Participants) | 22 | 22
  Week 9 | -5.1 (10.7) | -2.6 (7.6)
  Week 11: number analyzed (Participants) | 22 | 20
  Week 11 | -1.5 (12.5) | -1.6 (6.1)
  Week 13: number analyzed (Participants) | 23 | 22
  Week 13 | -2.0 (11.3) | -1.0 (10.0)
  Week15: number analyzed (Participants) | 4 | 13
  Week15 | -7.5 (5.1) | -2.3 (6.2)
  Week 17: number analyzed (Participants) | 4 | 9
  Week 17 | -7.3 (12.7) | -7.7 (12.2)
  Week 19: number analyzed (Participants) | 4 | 9
  Week 19 | -8.0 (8.4) | 0.4 (10.7)
  Week 21: number analyzed (Participants) | 4 | 9
  Week 21 | -8.0 (16.4) | -5.8 (10.1)
  Week 23: number analyzed (Participants) | 4 | 9
  Week 23 | 1.0 (9.0) | -3.6 (8.2)
  Week 25: number analyzed (Participants) | 4 | 16
  Week 25 | -9.0 (13.2) | -2.6 (11.2)
  Week 27: number analyzed (Participants) | 4 | 16
  Week 27 | -3.0 (10.4) | 3.5 (10.5)
  Week 29: number analyzed (Participants) | 4 | 16
  Week 29 | -8.3 (8.4) | 0.4 (11.2)
  Week 33: number analyzed (Participants) | 4 | 16
  Week 33 | -12.0 (20.7) | 4.6 (8.9)

6. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Change from baseline in pulse rate and at baseline values were reported for this outcome measure.
Time Frame: Baseline, Change at Weeks 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 33
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Beats per minute
  Baseline | 74.1 (11.8) | 74.2 (11.0)
  Week 2 | 2.1 (9.6) | 0.6 (6.9)
  Week 3: number analyzed (Participants) | 23 | 23
  Week 3 | -0.6 (8.0) | -1.1 (6.0)
  Week 5: number analyzed (Participants) | 22 | 23
  Week 5 | 0.0 (7.3) | -0.3 (8.0)
  Week 7: number analyzed (Participants) | 23 | 22
  Week 7 | -0.3 (9.2) | 0.0 (7.9)
  Week 9: number analyzed (Participants) | 22 | 22
  Week 9 | -1.0 (11.1) | 1.5 (9.0)
  Week 11: number analyzed (Participants) | 22 | 20
  Week 11 | -1.7 (10.8) | 0.6 (6.6)
  Week 13: number analyzed (Participants) | 23 | 22
  Week 13 | 3.3 (11.9) | 0.5 (6.9)
  Week15: number analyzed (Participants) | 4 | 13
  Week15 | -5.8 (10.4) | 5.0 (10.1)
  Week 17: number analyzed (Participants) | 4 | 9
  Week 17 | -6.3 (8.8) | -2.2 (5.0)
  Week 19: number analyzed (Participants) | 4 | 9
  Week 19 | -3.5 (13.7) | 2.9 (6.5)
  Week 21: number analyzed (Participants) | 4 | 9
  Week 21 | -5.5 (12.8) | -1.6 (5.0)
  Week 23: number analyzed (Participants) | 4 | 9
  Week 23 | -3.3 (10.5) | -3.1 (9.0)
  Week 25: number analyzed (Participants) | 4 | 16
  Week 25 | -6.3 (12.5) | 1.8 (7.6)
  Week 27: number analyzed (Participants) | 4 | 16
  Week 27 | -0.8 (16.0) | 2.9 (7.2)
  Week 29: number analyzed (Participants) | 4 | 16
  Week 29 | 2.5 (14.8) | 5.9 (8.8)
  Week 33: number analyzed (Participants) | 4 | 16
  Week 33 | -0.5 (15.3) | 6.2 (10.0)

7. Secondary Outcome: Change From Baseline in Body Temperature
Description: Change from baseline in body temperature and at baseline values were reported for this outcome measure.
Time Frame: Baseline, Change at Weeks 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 33
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Degree Celsius
  Baseline | 36.4 (0.4) | 36.6 (0.2)
  Week 2 | 0.1 (0.4) | -0.0 (0.3)
  Week 3: number analyzed (Participants) | 23 | 23
  Week 3 | 0.0 (0.2) | -0.1 (0.3)
  Week 5: number analyzed (Participants) | 22 | 23
  Week 5 | 0.0 (0.4) | -0.1 (0.3)
  Week 7: number analyzed (Participants) | 23 | 22
  Week 7 | 0.1 (0.3) | -0.0 (0.3)
  Week 9: number analyzed (Participants) | 22 | 22
  Week 9 | 0.0 (0.4) | -0.1 (0.3)
  Week 11: number analyzed (Participants) | 22 | 20
  Week 11 | 0.1 (0.3) | -0.0 (0.3)
  Week 13: number analyzed (Participants) | 23 | 22
  Week 13 | -0.1 (0.4) | -0.0 (0.2)
  Week 15: number analyzed (Participants) | 4 | 13
  Week 15 | 0.2 (0.2) | 0.1 (0.2)
  Week 17: number analyzed (Participants) | 4 | 9
  Week 17 | 0.1 (0.2) | 0.1 (0.2)
  Week 19: number analyzed (Participants) | 4 | 9
  Week 19 | 0.1 (0.4) | 0.1 (0.3)
  Week 21: number analyzed (Participants) | 4 | 9
  Week 21 | -0.0 (0.1) | -0.1 (0.5)
  Week 23: number analyzed (Participants) | 4 | 9
  Week 23 | 0.2 (0.2) | 0.0 (0.3)
  Week 25: number analyzed (Participants) | 4 | 16
  Week 25 | 0.1 (0.2) | 0.0 (0.2)
  Week 27: number analyzed (Participants) | 4 | 16
  Week 27 | 0.1 (0.1) | 0.1 (0.2)
  Week 29: number analyzed (Participants) | 4 | 16
  Week 29 | 0.1 (0.3) | -0.1 (0.4)
  Week 33: number analyzed (Participants) | 4 | 16
  Week 33 | 0.1 (0.1) | -0.1 (0.3)

8. Secondary Outcome: Number of Participants With Abnormalities in Electrocardiogram (ECG)
Description: ECG abnormalities criteria included: 1) QTc interval adjusted according to Bazett formula (QTcB) in millisecond (msec): greater than (>) 450, >480, >500, increase from baseline >30, increase from baseline >60; 2) QTc interval adjusted according to Fridericia formula (QTcF) (msec): >450, >480, >500, increase from baseline >30, increase from baseline >60; 3) Heart rate (bpm): RR decrease >25% and to a VR (interval between QRS wave and T wave on ECG) >100; RR (interval between 2 successive R waves on ECG) increase >25% and to a VR <50; 4) Pulse rate (msec): increase >25% and to a value >200; 5) QT (msec): >450, >480, >500, increase from baseline >30, increase from baseline >60; 6) QRS (msec): increase >25% and to a value >110. Categories (timepoints) with at least 1 participant having ECG abnormality in any of the reporting arms, were reported for this outcome measure.
Time Frame: Weeks 3, 7, 11, 13, 17, 21, 25, 33
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Participants
  Week 3 (Not Clinically Significant) | 3 | 4
  Week 3 (Clinically Significant): number analyzed (Participants) | 23 | 23
  Week 3 (Clinically Significant) | 1 | 0
  Week 7 (Not Clinically Significant): number analyzed (Participants) | 22 | 22
  Week 7 (Not Clinically Significant) | 3 | 4
  Week 7 (Clinically Significant): number analyzed (Participants) | 22 | 22
  Week 7 (Clinically Significant) | 0 | 0
  Week 11 (Not Clinically Significant): number analyzed (Participants) | 22 | 20
  Week 11 (Not Clinically Significant) | 4 | 4
  Week 11 (Clinically Significant): number analyzed (Participants) | 22 | 20
  Week 11 (Clinically Significant) | 1 | 0
  Week 13 (Not Clinically Significant): number analyzed (Participants) | 23 | 22
  Week 13 (Not Clinically Significant) | 6 | 4
  Week 13 (Clinically Significant): number analyzed (Participants) | 23 | 22
  Week 13 (Clinically Significant) | 1 | 0
  Week 17 (Not Clinically Significant): number analyzed (Participants) | 4 | 9
  Week 17 (Not Clinically Significant) | 0 | 0
  Week 17 (Clinically Significant): number analyzed (Participants) | 4 | 9
  Week 17 (Clinically Significant) | 0 | 0
  Week 21 (Not Clinically Significant): number analyzed (Participants) | 4 | 9
  Week 21 (Not Clinically Significant) | 1 | 1
  Week 21 (Clinically Significant): number analyzed (Participants) | 4 | 9
  Week 21 (Clinically Significant) | 0 | 0
  Week 25 (Not Clinically Significant): number analyzed (Participants) | 4 | 16
  Week 25 (Not Clinically Significant) | 1 | 1
  Week 25 (Clinically Significant): number analyzed (Participants) | 4 | 16
  Week 25 (Clinically Significant) | 0 | 0
  Week 33 (Not Clinically Significant): number analyzed (Participants) | 3 | 16
  Week 33 (Not Clinically Significant) | 0 | 2
  Week 33 (Clinically Significant): number analyzed (Participants) | 3 | 16
  Week 33 (Clinically Significant) | 0 | 0

9. Secondary Outcome: Percentage Change From Baseline in Urinary Protein to Creatinine Ratio (UPCR) at Weeks 2, 5, 9 and 13
Description: UPCR is a ratio between two measured substances in urine: mmol of creatinine, reported in units mg/mmol. A decrease in UPCR may be associated with improved renal and cardiovascular function.
Time Frame: Baseline, Weeks 2, 5, 9 and 13
Population: FAS was defined as all enrolled subjects who had received at least one dose of study treatment and had at least one post-baseline measurement of UPCR based on 24-hour urine collected. Here, 'Number Analyzed' signifies number of participants evaluable for the specific timepoints.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Percent change
  Week 2: number analyzed (Participants) | 0 | 0
  Week 5: number analyzed (Participants) | 20 | 20
  Week 5 | 6.250 [-7.035 to 21.433] | -3.788 [-11.344 to 4.411]
  Week 9: number analyzed (Participants) | 19 | 20
  Week 9 | -11.335 [-20.746 to -0.807] | -2.354 [-11.069 to 7.215]
  Week 13: number analyzed (Participants) | 21 | 19
  Week 13 | -12.283 [-26.096 to 4.112] | -0.045 [-9.528 to 10.432]

10. Secondary Outcome: Percentage Change From Baseline in Estimated Glomerular Filtration Rate (eGFR ) at Weeks 3, 5, 9 and 13
Description: The eGFR was calculated using 4 variable formula developed by the modification of diet in renal disease (MDRD) study group. The 4 variables needed to estimate glomerular filtration rate (GFR) using this formula were serum creatinine concentration, age, sex (for females, eGFR was multiplied by 0.742) and ethnic origin (for African-Caribbean people only, eGFR was multiplied by 1.212). Thus eGFR in milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) = 175*(sCr/88.4)^-1.154*(Age)^-0.203*(0.742 if female)*(1.212 if African-Caribbean). Baseline eGFR was determined predose at Week 0 (Day 1). For Baseline eGFR, the "Low eGFR" group was defined as baseline eGFR < 45 mL/min/1.73m2, and the "High eGFR" group was defined as baseline eGFR > 45 mL/min/1.73 m2.
Time Frame: Baseline, Weeks 3, 5, 9 and 13
Population: as for outcome 9
Measure: Least Squares Mean (90% Confidence Interval); unit: Percent change
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Percent change
  Week 3: number analyzed (Participants) | 23 | 22
  Week 3 | 5.657 [-0.722 to 12.446] | -0.180 [-4.179 to 3.987]
  Week 5: number analyzed (Participants) | 21 | 23
  Week 5 | 2.174 [-3.012 to 7.637] | -2.038 [-8.008 to 4.319]
  Week 9: number analyzed (Participants) | 22 | 22
  Week 9 | -1.536 [-15.575 to 14.838] | -5.017 [-11.596 to 2.052]
  Week 13: number analyzed (Participants) | 23 | 22
  Week 13 | 2.892 [-6.096 to 12.740] | -12.217 [-18.831 to -5.063]

11. Secondary Outcome: Serum PF-06730512 Concentration Versus Time Summary
Time Frame: For 12-Week treatment(WT):pre-dose on Day1,8,15,29,43,57,71,follow-up(Fup)visit on Day85,99,113,141,For 24-WT:pre-dose on Day1,8,15,29,43,57,71,85,99,113,127,141,155,Fup visit on Day169,183,197,225;1hour post-dose on Day1,71,155(only applicable for 24-WT)
Population: The PK concentration analysis set was defined as all enrolled participants treated who received at least one dose of PF-06730512 and had at least 1 measurable concentration. Here, 'Number Analyzed' signifies number of participants evaluable for the specific rows.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Microgram per milliliter
  Day 1: Pre-dose (12,24WT): number analyzed (Participants) | 19 | 24
  Day 1: Pre-dose (12,24WT) | 0 (0) | 0 (0)
  Day 1: Post-dose (12,24WT): number analyzed (Participants) | 17 | 22
  Day 1: Post-dose (12,24WT) | 279.4 (86.548) | 71.94 (29.668)
  Day 8: Pre-dose (12,24WT): number analyzed (Participants) | 1 | 10
  Day 8: Pre-dose (12,24WT) | 39.50 (NA) — Standard deviation could not be estimated as only one participant was evaluated. | 13.09 (6.9363)
  Day 15: Pre-dose (12,24WT): number analyzed (Participants) | 23 | 21
  Day 15: Pre-dose (12,24WT) | 16.45 (11.266) | 5.096 (3.1184)
  Day 29: Pre-dose (12,24WT): number analyzed (Participants) | 21 | 19
  Day 29: Pre-dose (12,24WT) | 24.92 (20.256) | 6.916 (5.0154)
  Day 43: Pre-dose (12,24WT): number analyzed (Participants) | 20 | 19
  Day 43: Pre-dose (12,24WT) | 29.96 (22.062) | 6.991 (5.5862)
  Day 57: Pre-dose (12,24WT): number analyzed (Participants) | 21 | 18
  Day 57: Pre-dose (12,24WT) | 32.56 (23.031) | 7.664 (6.1325)
  Day 71: Pre-dose (12,24WT): number analyzed (Participants) | 17 | 17
  Day 71: Pre-dose (12,24WT) | 27.32 (16.688) | 6.736 (5.6237)
  Day 71: Post-dose(12,24WT): number analyzed (Participants) | 20 | 17
  Day 71: Post-dose(12,24WT) | 298.6 (208.87) | 129.2 (201.50)
  Day 85: Pre-dose (24WT): number analyzed (Participants) | 4 | 13
  Day 85: Pre-dose (24WT) | 41.15 (23.516) | 7.597 (6.9184)
  Day 85/Fup (12 WT): number analyzed (Participants) | 19 | 7
  Day 85/Fup (12 WT) | 27.19 (21.589) | 6.884 (7.1511)
  Day 99/Fup (12 WT): number analyzed (Participants) | 19 | 7
  Day 99/Fup (12 WT) | 11.50 (12.948) | 2.313 (3.1827)
  Day 113/Fup (12 WT): number analyzed (Participants) | 19 | 7
  Day 113/Fup (12 WT) | 4.991 (6.1121) | 0.6356 (0.81118)
  Day 141/Fup (12 WT): number analyzed (Participants) | 18 | 7
  Day 141/Fup (12 WT) | 1.385 (2.1196) | 0.1438 (0.21666)
  Day 99: Pre-dose (24WT): number analyzed (Participants) | 4 | 9
  Day 99: Pre-dose (24WT) | 35.65 (16.065) | 7.084 (6.9224)
  Day 113: Pre-dose (24WT): number analyzed (Participants) | 4 | 6
  Day 113: Pre-dose (24WT) | 42.40 (25.049) | 9.442 (8.6965)
  Day 127: Pre-dose (24WT): number analyzed (Participants) | 3 | 6
  Day 127: Pre-dose (24WT) | 30.67 (5.3463) | 6.732 (5.2295)
  Day 141: Pre-dose (24WT): number analyzed (Participants) | 4 | 7
  Day 141: Pre-dose (24WT) | 38.00 (13.880) | 8.957 (10.753)
  Day 155: Pre-dose (24WT): number analyzed (Participants) | 3 | 8
  Day 155: Pre-dose (24WT) | 32.57 (5.8287) | 7.585 (8.1601)
  Day 155: Post-dose (24WT): number analyzed (Participants) | 4 | 8
  Day 155: Post-dose (24WT) | 313.3 (63.793) | 62.71 (41.324)
  Day 169: Pre-dose/Fup (24WT): number analyzed (Participants) | 4 | 16
  Day 169: Pre-dose/Fup (24WT) | 29.32 (15.338) | 7.989 (7.4740)
  Day 183/Fup (24WT): number analyzed (Participants) | 4 | 16
  Day 183/Fup (24WT) | 25.79 (30.417) | 3.046 (3.8895)
  Day 197/Fup (24WT): number analyzed (Participants) | 4 | 16
  Day 197/Fup (24WT) | 6.108 (4.0049) | 1.048 (1.4978)
  Day 225/Fup (24WT): number analyzed (Participants) | 4 | 16
  Day 225/Fup (24WT) | 2.009 (1.6808) | 0.2659 (0.45714)

12. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibody(NAb)
Description: Number of participants with positive ADA and/or NAb were reported for this outcome measure.
Time Frame: From Day 1 of treatment up to Week 33
Population: The immunogenicity analysis population included all treated participants with at least 1 ADA sample (pre-dose or post-treatment) analyzed. Participants those had only pre-dose baseline data and no post-treatment immunogenicity data, was not evaluated for subject-level ADA and NAb status. Here, 'Number Analyzed' signifies number of participants evaluable for the specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
Number analyzed (Participants) | 23 | 24
Participants
  ADA Positive | 1 | 0
  nAb Positive | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 of treatment up to 9 weeks after last dose of study treatment (up to Week 33)
Description: Same event may appear as both non-SAE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participants, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-06730512 1000 mg IV | PF-06730512 300 mg IV
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 2/23 | 2/24
Other Adverse Events (participants affected / at risk) | 11/23 | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06730512 1000 mg IV (N=23) | PF-06730512 300 mg IV (N=24)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06730512 1000 mg IV (N=23) | PF-06730512 300 mg IV (N=24)
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 3 | 2
Oedema (General disorders) | 0 | 2
Pyrexia (General disorders) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
SARS-CoV-2 test positive (Investigations) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT03448692/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT03448692/SAP_001.pdf